CLINICAL TRIAL: NCT01225757
Title: Comparison of Traditional (Central Venous Pressure (CVP) and Urine Output Guided) Versus Echocardiography Guided Fluid Management in Patients Undergoing Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Brief Title: Comparison of Traditional and Echocardiography Guided Fluid Management During Cytoreductive Surgery With HIPEC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical problems prior to the recruitment phase
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0168-10-FB
Record Dates: First submitted 2010-07-14; First posted 2010-10-21 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Peritoneal Neoplasms; Echocardiography Guided Fluid Management
Keywords: Echocardiography; HIPEC
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Echocardiography (Experimental): These patients will have echocardiography guided fluid management
  Interventions: Device: Echocardiogram
- Traditional fluid management (Active Comparator): Fluid management will be guided by monitoring of central venous pressure and urine output.
  Interventions: Device: Echocardiogram

INTERVENTIONS:
Device: Echocardiogram — Echocardiography will be utilized during the procedure to guide fluid management.
  Other Names: Phillips Echocardiography machines

SUMMARY:
Cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (HIPEC) is performed in patients with peritoneal tumors. Classically, this procedure is prolonged in duration and involves significant fluid shifts. Patients receive a large amount of volume replacement during this procedure (between 10 and 20 liters). The traditional methods to monitor adequacy of volume replacement are measurement of urine output and central venous pressure. There are drawbacks of any method of intravascular volume status measurement which may lead to over or under replacement of fluids. If fluid replacement is underestimated, the patient may suffer from adverse effects such as hypotension and renal dysfunction. However, the excessive administration of fluids may lead to other adverse events, including cardiac dysrhythmias and heart failure. The hypothesis of this study is that patients in whom volume status is maintained by utilizing a transesophageal echocardiogram will have better maintenance of fluid status while avoiding intravascular volume overload.

DETAILED DESCRIPTION:
Cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (HIPEC) is a procedure in which peritoneal surface tumors are removed followed by infusion of a heated chemotherapeutic solution into the abdominal cavity. This procedure is typically 6-10 hours in duration and is accompanied by significant fluid shifts and hemodynamic changes. Patients frequently receive between 10 and 20 liters of fluid during the procedure. Patients undergoing cytoreductive surgery with HIPEC also experience vasodilatation and a hyperdynamic cardiac state during the hyperthermic period. Classically, the need for volume replacement has been guided by following a patient's urine output (UOP) and the use of central venous pressure (CVP). However, several studies have shown that CVP is not a reliable measure of intravascular fluid status.

We hypothesize that patients undergoing echocardiography guided anesthesia management (EGAM) will receive significantly less fluid during the operative period when compared to more traditional fluid therapy guided by monitoring of urine output and central venous pressure. In addition to the primary endpoint of a decrease in fluid administration, we would predict a decrease in time to extubation, intensive care unit length of stay, hospital length of stay, post operative oxygen requirements, post operative complications including tachyarrhythmias, heart failure and pulmonary edema, and length of time to recovery of bowel function.

Patients presenting for cytoreductive surgery with HIPEC will be randomized into one of two groups, the echocardiography guided fluid management group or the traditional CVP/UOP fluid guided group. For patients in the echocardiography arm, this monitor will be used to optimize preload, contractility, heart rate and cardiac output. Patients in the CVP/UOP arm will receive the current standard of fluid administration to maintain adequate urine output. All patients presenting for the procedure will be offered an opportunity for admission into the study. Exclusion criteria include any absolute contraindications to transesophageal echocardiography, including cervical spine instability, esophageal strictures, webs or rings, patient refusal, esophageal perforation, obstructive esophageal neoplasms (Savage 2004).

A follow-up evaluation will be completed during the remainder of the patient's hospitalization to evaluate the previously discussed endpoints. The goal is to determine the optimal fluid management strategy to decrease morbidity in the post-operative period in patients undergoing cytoreductive surgery with hyperthermic intraperitoneal chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing cytoreductive surgery with hyperthermic intraperitoneal chemotherapy who are 19 years of age and older will be eligible for inclusion in this study.

Exclusion Criteria:

* Inability to give informed consent
* Absolute contraindications to transesophageal echocardiography, including cervical spine instability, esophageal strictures, webs or rings, patient refusal, esophageal perforation, obstructive esophageal neoplasms.
* Relative contraindications to transesophageal echocardiography esophageal diverticulum, large hiatal hernias, recent esophageal or gastric surgery, esophageal varices, history of dysphagia or odynophagia, cervical arthritis, history of radiation to the mediastinum, deformities of the oral pharynx and severe coagulopathy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11 (Estimated); Primary Completion 2011-08-31 (Actual); Study Completion 2011-08-31 (Actual)

PRIMARY OUTCOMES:
Fluid administration decrease | One day (intraoperative period)
  The amount of fluid administered during the intraoperative period will be monitored and recorded. The outcome measure of interest is the difference between fluid given in the standard group vs the echo guided fluid management group.

SECONDARY OUTCOMES:
Time to extubation | An average of up to two weeks
  The amount of time for participants to be extubated
Intensive care unit and hospital length of stay | An average of up to two weeks
  Duration of stay in intensive care and overall time in hospital
Post operative oxygen requirements | An average of up to two weeks
  The need, level and duration of any required post-operative oxygen
Cardiac complications | An average of up to two weeks
  Post operative cardiac complications including tachyarrhythmias, heart failure and pulmonary edema

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Duhachek-Stapelman, MD, Principal Investigator — University of Nebraska